CLINICAL TRIAL: NCT00501709
Title: Prevention of Autoimmune Destruction and Rejection of Human Pancreatic Islets Following Transplantation for Insulin Dependent Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39-42C
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Abatacept; efalizumab; Immunosuppressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Allogenic pancreatic islet transplant using belatacept and raptiva
  Interventions: Drug: Belatacept and Raptiva

INTERVENTIONS:
Drug: Belatacept and Raptiva — immunosuppressant agent to prevent rejection in transplant recipients
  Other Names: immunosuppressant

SUMMARY:
Pancreatic islets are the part of the pancreas that produce insulin and help control the blood sugar. This study aims to improve islet transplantation as a treatment for Type 1 Diabetes by using a new combination of immunosuppressive drugs that have been successful in treating other autoimmune diseases and in preventing kidney transplant rejection.

DETAILED DESCRIPTION:
The primary objective of these studies is to assess the efficacy and safety of allogeneic pancreatic islet transplantation in the treatment of type I diabetes mellitus. A secondary study objective is to evaluate the efficacy of various immunosuppressive protocols and agents in preventing autoimmune destruction and rejection of allogeneic islet transplants. A tertiary objective is to determine the safety and efficacy of allogeneic pancreatic islet transplantation in patients who have received another organ transplant such as a kidney or liver.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* Metabolic lability/instability characterized by hypoglycemia or ketoacidosis(>2 hospital admissions in the previous year), erratic glucose profiles(MAGE >120mg/dL), or disruption in lifestyle(danger to life, self or others). Reduced awareness of hypoglycemia or > 1 episode in the last 1.5 years of severe hypoglycemia.
* Persistently poor glucose control (as defined by HgbA1c>10% at the end of six months of intensive management efforts with diabetes care team.
* Progressive secondary complications as defined by

  * a new diagnosis by an ophthalmologist of proliferative retinopathy or clinically significant macular edema or therapy with photocoagulation during the last year; or
  * urinary albumin excretion rate >300mg/day but proteinuria <3g/day; or
  * symptomatic autonomic neuropathy (as defined by postural hypotension in the setting of euvolemia, gastroparesis or diarrhea attributed to diabetic neuropathy, or neuropathic bladder as diagnosed by an urologist)

Exclusion Criteria:

* Patient weighs more than 80kg or body mass index BMI>28
* Patient's insulin requirement is >55 Units/day.
* Current use of immunosuppressive agents.
* History of malignancy within 10 years (except for adequately treated basal or squamous cell CA of the skin).
* Active peptic ulcer disease.
* Severe unremitting diarrhea or other GI disorders potentially interfering with the ability to absorb oral medications.
* Untreated proliferative retinopathy.
* Pregnancy or breastfeeding.
* Female subjects not post-menopausal or surgically sterile, or not using an acceptable method or contraception.
* Active infections.
* Major ongoing psychiatric illness.
* Ongoing substance abuse, drug or alcohol; or recent history of noncompliance.
* Portal hypertension or history of significant liver disease.
* Lymphopenia (<1000/ul) or leukopenia (<3000 total leukocytes/ul) or an absolute CD4 count <500/ul.
* Presence or history of panel-reactive anti-HLA antibody >20%.
* Evidence of acute EBV infection (IgM>IgG) OR no serologic evidence of previous exposure to EBV (IgG>IgM).
* Serologic evidence of infection with HIV or HbsAg or HCV Ab positive.
* Creatinine clearance <60ml/min/m2.
* Positive lymphocytoxic cross-match using donor lymphocytes and serum

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
lnsulin independence | monthly
  improved glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Stock, M.D., Ph.D., Principal Investigator — University of California, San Francisco; Andrew Posselt, M.D., Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States